CLINICAL TRIAL: NCT00811785
Title: Molecular Bases of Response to Copper Treatment in Menkes Disease, Related Phenotypes, and Unexplained Copper Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cyprium Therapeutics, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090059; 09-CH-0059
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2019-08

CONDITIONS: Menkes Disease; Occipital Horn Syndrome; Unexplained Copper Deficiency
Keywords: Copper Deficiency; Menkes Disease; Neurodegeneration; Occipital Horn Syndrome; Copper
MeSH Terms: conditions — Menkes Kinky Hair Syndrome; Occipital horn syndrome; Nerve Degeneration | interventions — copper histidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Copper Histidine — Daily subcutaneous injections for three years

SUMMARY:
Menkes disease and occipital horn syndrome are two forms of copper deficiency that must be diagnosed and treated very early in life to prevent serious developmental problems. However, these and other forms of copper deficiency are not very well understood, and further research is needed to determine whether certain treatments are useful in treating copper deficiency. One such treatment is copper histidine, a copper replacement that can be injected directly into the body to avoid absorption through the gastrointestinal tract. This study will investigate the effectiveness, side effects, and dosage of copper histidine treatment for patients with copper deficiency. It will also collect medical history information from patients to allow researchers to study possible genetic and nongenetic origins of copper deficiency.

This study will include 100 subjects, all of whom will be children and adults who have been diagnosed with Menkes disease, occipital horn syndrome, or other unexplained copper deficiency.

Patients will receive a prescribed dose of copper histidine, which will be administered daily as an injection.

During the study, patients will be admitted to the NIH Clinical Center on an outpatient basis to evaluate their response to the copper histidine treatment. These evaluations will take place every 8 months, with a final evaluation performed after 3 years of treatment. During the outpatient visits, patients will be required to give blood and urine samples for testing and undergo ultrasound testing. They will also undergo brain MRI scans at the initial visit and at the 16-month and 36-month visits. Patients who agree will give additional blood samples for genetic research purposes.

DETAILED DESCRIPTION:
Study Description:

The purpose of this study is to allow currently enrolled participants to complete their three-year course of subcutaneous Copper Histidinate treatment under the protocol. We hypothesize that subcutaneous injections of this drug will raise serum copper levels and ceruloplasmin levels in enrolled participants, improve neurodevelopmental and neurological outcomes, and reduce mortality compared to untreated affected subjects.

Objectives:

-Primary Objective: Evaluate responses to Copper Histidinate treatment for clinical care.

Endpoints:

-Completion of three years treatment by 13 remaining subjects

Study Population:

The 13 remaining subjects

Phase: Clinical Care/Treatment only

Description of Sites/Facilities Enrolling Participants: The study will occur at the NIH Clinical Center

Description of Study Intervention:

The study intervention is administration of Copper Histidinate in dose(s) prescribed as follows: 250 microgram sc b.i.d. in infants up to 12 months of age, and 250 microgram sc q.d. for infants and children older than 12 months. The total duration of copper histidinate treatment will not exceed three years.

Study Duration:

The estimated time from when the study opens to enrollment until completion is approximately 151 months (02/27/2009-09/30/2021). (May end sooner pending FDA new drug approval.)

Participant Duration:

The time it will take for each individual participant to complete all participant visits is approximately 36 months. There are 13 subjects with a total of 31 visits to complete.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form by parent or legal guardian, or the subject himself/herself.
2. Male or female, aged 0 to 80 years.
3. Diagnosed with classic Menkes disease, Occipital Horn Syndrome (OHS), or unexplained copper deficiency.
4. Serum copper level results between 0 and 75 mg/dl (normal range 80-180 microgram/dl).
5. Ability to adhere to the prescribed subcutaneous Copper Histidinate injection regimen.
6. Willingness to comply with all study visits and procedures.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pre-existing liver (e.g., hepatitis, biliary atresia, cirrhosis) or kidney disease (e.g., serum creatinine >1.0 mg/dL)
2. History of bleeding diatheses
3. Pregnancy or lactation
4. Diagnosis of Wilson disease
5. Any disease or condition that, in the opinion of the Investigator, has a high probability of precluding the patient from completing the study or where the patient cannot or will not appropriately comply with study requirements
6. Participation in any other investigational trial in which receipt of investigational drug or device occurred within 30 days prior to screening for this study
7. History of diagnosed drug or alcohol dependence within the previous 3 years
8. Any disease process that may adversely affect gastrointestinal absorption, e.g. celiac sprue
9. Chronic/severe cardiac disease (applies to adult subjects only) that could make participating in a clinical trial physically demanding, including but not limited to cardiac insufficiency, arrhythmias, bradycardia, or hypotension, unless associated with other features of dysautonomia, as in OHS.
10. History of cerebrovascular accident (applies to adult subjects only) that could make participating in a clinical trial difficult for the subject.

Adults who are, or who may be, unable to consent will not be allowed to participate in this study. This is because we did not encounter subjects in this category for whom enrollment would be necessary or appropriate in our previous studies (90-CH-0149, 90-N-0149) with this IND. The main populations to be recruited are 1) pediatric subjects under 18 years of age with inherited copper transport disorders, and 2) non-cognitively-impaired adults with unexplained copper deficiency.

NIH employees are eligible to participate in this protocol if they meet the Inclusion criteria and have no exclusion criteria. Recruitment, enrollment and compensation of NIH employee subjects will be consistent with the Guidelines for the Inclusion of Employees in NIH Intramural Research Studies (December 2015) and NIH Policy Manual Chapter 2300-630-3, "Leave Policy for NIH Employees Participating in NIH Medical Research Studies". The consenting research team member will make the NIH Information Sheet on Employee Research Participation available to staff members who are considering enrolling.

If the individual requesting to participate in the protocol is a co-worker, the consent from the NIH staff member (co-worker) will not be obtained by the staff member s direct supervisor but by another research staff member approved for obtaining informed consent who is not a co-worker.

Neither participation nor refusal to participate as a subject in this protocol will have an effect, either beneficial or adverse, on the participant s employment or position at NIH.

Employee subjects' privacy and confidentiality will be respected by protocol and consenting staff the same as for all subjects participating in research protocols. However, all subjects will be made aware that there are limits to these protections.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-02-27; Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
To assess neurological improvement in patients with OHS or unexplained copper deficiency treated with subcutaneous CuHis injections. | Three years
  Neurological Improvement: reduction in dysautonomia symptoms in OHS, and improved nerve conduction tests in unexplained copper deficiency

SECONDARY OUTCOMES:
To assess survival in classic Menkes disease subjects treated with subcutaneous CuHis injections in comparison with classic Menkes patients who did not receive any type of copper treatment. | Continuously
  Under-three Mortality. This endpoint will be assessed continuously

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kaler SG, Goldstein DS, Holmes C, Salerno JA, Gahl WA. Plasma and cerebrospinal fluid neurochemical pattern in Menkes disease. Ann Neurol. 1993 Feb;33(2):171-5. doi: 10.1002/ana.410330206. PMID 8434878
- [Background] Kaler SG, Westman JA, Bernes SM, Elsayed AM, Bowe CM, Freeman KL, Wu CD, Wallach MT. Gastrointestinal hemorrhage associated with gastric polyps in Menkes disease. J Pediatr. 1993 Jan;122(1):93-5. doi: 10.1016/s0022-3476(05)83496-1. PMID 8419622
- [Background] Kaler SG, Gahl WA, Berry SA, Holmes CS, Goldstein DS. Predictive value of plasma catecholamine levels in neonatal detection of Menkes disease. J Inherit Metab Dis. 1993;16(5):907-8. doi: 10.1007/BF00714295. No abstract available. PMID 8295415
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-CH-0059.html